CLINICAL TRIAL: NCT05907590
Title: Proprioception and Interoception in Patients With Fibromyalgia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: TRACE labs Ziekenhuis Oost-Limburg (ZOL) (Unknown)
Responsible Party: Principal Investigator, Indra Ramakers, PhD researcher, Hasselt University
Other Study IDs: B1152022000007
Record Dates: First submitted 2023-05-24; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Fibromyalgia
Keywords: Interoception; Proprioception; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Fibromyalgia: Patients with fibromyalgia diagnosed using the ACR criteria (American College of Rheumatology, Wolfe et al., 2010; 2016).
  Interventions: Other: Interoceptive accuracy measurement; Other: Interoceptive sensibility measurement; Other: Interoceptive awareness measurement; Other: Proprioceptive accuracy measurement during postural control; Other: Proprioceptive accuracy measurement of the neck
- Healthy Controls: Healthy controls will consist of people who experience few physical complaints in daily life. The healthy controls will thus be screened for inclusion using the CSD (Checklist for Symptoms in Daily life; Walentynowicz, et al., 2018). Only volunteers with a score of 75 or lower on this questionnaire will be included
  Interventions: Other: Interoceptive accuracy measurement; Other: Interoceptive sensibility measurement; Other: Interoceptive awareness measurement; Other: Proprioceptive accuracy measurement during postural control; Other: Proprioceptive accuracy measurement of the neck

INTERVENTIONS:
Other: Interoceptive accuracy measurement — Interoceptive accuracy will be measured using the Respiratory Occlusion Discrimination Task (ROD task; Van Den Houte et al., 2021). The ROD task measures how good subjects are at distinguishing the lengths of short (max 620 milliseconds) inspiratory occlusions (or respiratory interruptions).
Other: Interoceptive sensibility measurement — Interoceptive sensibility will be measured using two self-report questionnaires, the Interoceptive Sensitivity and Attention Questionnaire (ISAQ; Bogaerts et al., 2022) and the the Three-domain Interoceptive Sensations Questionnaire (THISQ; Vlemincx et al., 2021)
Other: Interoceptive awareness measurement — Interoceptive awareness will be measures using a visual analogue scale (VAS)
Other: Proprioceptive accuracy measurement during postural control — The effect of muscle vibration on center of gravity displacement (center of pressure or COP) will be examined. Muscle vibration of the m. triceps surae ("ankle" muscles) and the lumbar multifidus ("back" muscles) (Johanson et al., 2011; Brumagne et al., 2008; Claeys et al., 2011; Cleays et al., 2015) will be used to examine the role of proprioception during postural control.
Other: Proprioceptive accuracy measurement of the neck — The head reposition accuracy task will be carried out to assess proprioceptive accuracy of the neck. The most commonly used procedure is the head repositioning accuracy to neutral head position (HRA-to-NHP), first described by Revel and colleagues (1991).

SUMMARY:
The goal of this observational study is to learn about interoception and proprioception in patients with fibromyalgia. The main questions it aims to answer are:

* Is there a significant difference in interoception between patients with fibromyalgia and healthy controls?
* Is there a significant difference in proprioception between patients with fibromyalgia and healthy controls?

The participants will perform:

* The respiratory occlusion discrimination task
* A postural control task where the effect of muscle vibration on center of gravity displacement is examined
* The head repositioning accuracy task

The participants will also fill out different questionnaires.

Researchers will compare healthy controls to see if there is a significant difference.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic widespread pain condition characterized by point tenderness, fatigue, sleep disturbance, cognitive complaints, and increasing somatic complaints. With this case-control study we want to emphasize the importance of an integrative psychophysiological model for fibromyalgia, in which interoception and proprioception are being investigated.

Interoception has been described in the literature as "the overall process of how the nervous system senses, integrates, stores and displays information about the state of the internal body". Theory suggests that interoception should be divided into three measurable constructs: interoceptive accuracy (objective accuracy in detecting internal bodily sensations), interoceptive sensitivity (the self-perceived tendency to be internally self-focused), and interoceptive awareness (metacognition about his/her own interoceptive accuracy). Proprioception on the other hand, is described as the sense of body position and movement.

The first measurement will take place in the lab of REVAL Hasselt University. First, informed consent will be signed before any data collection takes place. This part of the experiment will take approximately 30 minutes.

Two proprioception tasks will be performed consecutively. The effect of muscle vibration on centre of gravity displacement (center of pressure or COP) will be examined. Muscle vibration of the m. triceps surae ("ankle" muscles) and the lumbar multifidus ("back" muscles) will be used to examine the role of proprioception during postural control. The displacement (magnitude) of the COP during standing will be assessed with a force plate. The muscle vibration induces muscle extension illusions, so that, in order to maintain balance, the subject, by a compensatory mechanism, will send the COP to the opposite side when he or she effectively uses the proprioceptors (muscle spindles) of the vibrated muscle. The same task will be performed on both a stable and an unstable surface.

The head reposition accuracy task will be carried out to assess neck proprioception. The most commonly used procedure is the head repositioning accuracy to neutral head position (HRA-to-NHP). During this procedure, the subject sits against a backrest. The subject is blindfolded to exclude visual input and wears a helmet containing a beam of light directed at a target 90 cm in front of the subject. The subject is instructed to look straight ahead and memorize this position. At that point, the test leader will mark off this point on the target. Subject's head is turned at an angle by the subject (active). Test subject will hereafter have to actively move the head back to the initial position. The direction of movement used are rotations, both to the left and to the right.

The second part of the experiment will take place in the TRACE labs of Ziekenhuis Oost Limburg (ZOL). It will take approximately 30 minutes. Participants will start with the interoceptive accuracy task using the Respiratory Occlusion Discrimination Task (ROD task). The ROD task measures how good subjects are at distinguishing the lengths of short (max 620 milliseconds) inspiratory occlusions (or respiratory interruptions). Occlusions of these lengths are not aversive or unpleasant. One trial consists of two occlusions within one inspiration (inter-occlusion interval = 300 milliseconds), one occlusion being the reference occlusion (always 440 milliseconds) and one occlusion being the test occlusion (longer or shorter than 440 milliseconds), administered in random order. The participant is asked to indicate which of the two occlusions was longest. An adaptive staircase paradigm is thus used to determine the just noticeable difference in lengths of inspiratory occlusions. The length of the task depends on the performance of the subject, but is on average 56 trials (= 15 minutes). After the experiment, another short side experiment of 16 trials will be conducted in which the participant should indicate how confident they were in their response on a Visual Analogue scale (VAS), in order to estimate interoceptive awareness. In the meantime, participants will be also asked to complete a questionnaire bundle at home (online), which takes approximately 45 minutes to complete.

The power calculations resulted in a total of 26 persons per group. Therefore the investigators plan to recruit a total of 52 people.

Primary outcomes are interoceptive accuracy, interoceptive sensibility, interoceptive awareness, and proprioceptive accuracy. Secondary outcome measures are psychological variables measured using questionnaires.

Descriptive statistics will be used to display baseline group characteristics. To evaluate between-group differences (i.e. the difference between patients with fibromyalgia and healthy controls regarding interoception, proprioception and psychological variables) t-tests will be used.

ELIGIBILITY:
Eligibility criteria healthy controls:

Inclusion Criteria:

Healthy controls will be selected so that there is an equal ratio between patients and healthy controls for

* Age group (per 5 years)
* Gender (including X)
* Educational attainment
* BMI

all participants need a score < 75 on the CSD (Walentynowicz et al., 2018)

Exclusion Criteria:

* Pregnancy
* Under the age of 18 or over the age of 65.
* Presence of a depressive episode, anxiety disorder, eating disorder, substance abuse, neurocognitive, or psychotic disorder diagnosed with DSM-V (Diagnostic and Statistical Manual of Mental Disorders; MINI-s; Overbeek et al., 1999).
* Presence of a chronic organic disorder (It is referred to as a chronic organic disorder if it has been present for a period of at least 3 months. Examples are: epilepsy, heart disease, rheumatism, asthma, diabetes, etc.) or acute organic disorder (fever, flu, etc.)
* Persistent physical complaints (e.g. hyperventilation complaints, long-term COVID, chronic pain or fatigue, chronic tinnitus, etc. )
* Neck complaints at the time of testing
* Recent whiplash trauma less than 3 months ago or more than 3 months ago with complaints still present
* Diagnosis of vestibular or neurological disorders
* Recent orthopedic problems of the lower extremities (e.g. acute ankle trauma) that may affect balance
* BMI>30

Eligibility criteria patients with fibromyalgia

Inclusion Criteria:

* Patients with fibromyalgia diagnosed using the ACR criteria (Wolfe et al., 2010; 2016).

Exclusion Criteria:

* Pregnancy
* Under the age of 18 or over the age of 65
* Primary depressive episode, anxiety disorder, eating disorder, substance abuse, neurocognitive, or psychotic disorder diagnosed with DSM-V (MINI-s; Overbeek et al., 1999).
* Presence of a chronic organic disorder (It is referred to as a chronic organic disorder if it has been present for a period of at least 3 months. Examples are: epilepsy, heart disease, rheumatism, asthma, diabetes, etc.) or acute organic disorder (fever, flu, etc.)
* Neck complaints at the time of testing (not related to the current problem)
* Recent whiplash trauma less than 3 months ago or more than 3 months ago with symptoms still present
* Diagnosis of organically explained vestibular or neurological disorders
* Recent orthopedic problems of the lower extremities (e.g., acute ankle trauma) that may affect balance
* BMI>30

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with fibromyalgia diagnosed according to the ACR criteria (Wolfe et al., 2010; 2016) are eligible to participate
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Interoceptive accuracy | 20 minutes
  Respiratory occlusion discrimination task (ROD task; Van Den Houte et al., 2021)
Interoceptive sensibility | 5 minutes
  Interoceptive Sensitivity and Attention Questionnaire (ISAQ; Bogaerts et al., 2022)
Interoceptive sensibility | 5 minutes
  THree-domain Interoceptive Sensations Questionnaire (THISQ; Vlemincx et al., 2021)
Interoceptive awareness | 5 minutes
  Visual analogue scale (0-100). A score of 0 indicates that participants are not certain at all of their answer, a score of 100 indicates that participants are entirely certain of their answer.
Proprioceptive accuracy | 5 minutes
  Head repositioning accuracy task
Proprioceptive accuracy | 30 minutes
  Postural control task

SECONDARY OUTCOMES:
Psychological variables | 5 minutes
  Checklist for Symptoms in Daily Life (CSD; Walentynowicz et al., 2018)
  Checklist for Symptoms in Daily Life (CSD; Walentynowicz et al., 2018)
  Checklist for Symptoms in Daily Life (CSD; Walentynowicz et al., 2018)
  Checklist for Symptoms in Daily Life (CSD; Walentynowicz et al., 2018)
Psychological variables | 5 minutes
  Positive and Negative Affect Scale (PANAS; Watson et al., 1988)
Psychological variables | 5 minutes
  Tellegen Absorption Scale (TAS; Tellegen & Atkinson, 1974)
Psychological variables | 10 minutes
  Traumatic Experiences Checklist (TEC; Nijenhuis et al., 2002)
Psychological variables | 5 minutes
  Toronto Alexithymia Scale (TAS-20; Bagby et al., 1994)
Psychological variables | 5 minutes
  Need for Controllability and Predictability Questionnaire (NCP-q; Ramakers et al., manuscript in preparation)
Psychological variables | 5 minutes
  Frost Multidimensional Perfectionism Scale (FMPS; Frost et al., 1990)
Psychological variables | 5 minutes
  Acceptance and Action Questionnaire-II (AAQ-II; Bond et al., 2011)

CONTACTS AND LOCATIONS:
Overall Officials: Katleen Bogaerts, PhD, Principal Investigator — Hasselt University
Locations (2):
- Belgium (2):
  - Hasselt University, Diepenbeek, Limburg
  - TRACE labs Ziekenhuis Oost-Limburg (ZOL), Lanaken, Limburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RL, Mease PJ, Russell AS, Russell IJ, Walitt B. 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria. Semin Arthritis Rheum. 2016 Dec;46(3):319-329. doi: 10.1016/j.semarthrit.2016.08.012. Epub 2016 Aug 30. PMID 27916278
- [Background] Khalsa SS, Adolphs R, Cameron OG, Critchley HD, Davenport PW, Feinstein JS, Feusner JD, Garfinkel SN, Lane RD, Mehling WE, Meuret AE, Nemeroff CB, Oppenheimer S, Petzschner FH, Pollatos O, Rhudy JL, Schramm LP, Simmons WK, Stein MB, Stephan KE, Van den Bergh O, Van Diest I, von Leupoldt A, Paulus MP; Interoception Summit 2016 participants. Interoception and Mental Health: A Roadmap. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Jun;3(6):501-513. doi: 10.1016/j.bpsc.2017.12.004. Epub 2017 Dec 28. PMID 29884281
- [Background] Garfinkel SN, Seth AK, Barrett AB, Suzuki K, Critchley HD. Knowing your own heart: distinguishing interoceptive accuracy from interoceptive awareness. Biol Psychol. 2015 Jan;104:65-74. doi: 10.1016/j.biopsycho.2014.11.004. Epub 2014 Nov 20. PMID 25451381
- [Background] Tuthill JC, Azim E. Proprioception. Curr Biol. 2018 Mar 5;28(5):R194-R203. doi: 10.1016/j.cub.2018.01.064. PMID 29510103
- [Background] Walentynowicz, M., Witthöft, M., Raes, F., Van Diest, I., & Van den Bergh, O. (2018). Sensory and affective components of symptom perception: a psychometric approach. Journal of Experimental Psychopathology, 9(2), 1-13. Doi: 10.5127/jep.059716
- [Background] Brumagne S, Janssens L, Knapen S, Claeys K, Suuden-Johanson E. Persons with recurrent low back pain exhibit a rigid postural control strategy. Eur Spine J. 2008 Sep;17(9):1177-84. doi: 10.1007/s00586-008-0709-7. Epub 2008 Jul 2. PMID 18594876
- [Background] Claeys K, Brumagne S, Dankaerts W, Kiers H, Janssens L. Decreased variability in postural control strategies in young people with non-specific low back pain is associated with altered proprioceptive reweighting. Eur J Appl Physiol. 2011 Jan;111(1):115-23. doi: 10.1007/s00421-010-1637-x. Epub 2010 Sep 8. PMID 20824281
- [Background] Claeys K, Dankaerts W, Janssens L, Pijnenburg M, Goossens N, Brumagne S. Young individuals with a more ankle-steered proprioceptive control strategy may develop mild non-specific low back pain. J Electromyogr Kinesiol. 2015 Apr;25(2):329-38. doi: 10.1016/j.jelekin.2014.10.013. Epub 2014 Oct 31. PMID 25467548
- [Background] Johanson E, Brumagne S, Janssens L, Pijnenburg M, Claeys K, Paasuke M. The effect of acute back muscle fatigue on postural control strategy in people with and without recurrent low back pain. Eur Spine J. 2011 Dec;20(12):2152-9. doi: 10.1007/s00586-011-1825-3. Epub 2011 May 1. PMID 21533851
- [Background] Cordo PJ, Gurfinkel VS, Brumagne S, Flores-Vieira C. Effect of slow, small movement on the vibration-evoked kinesthetic illusion. Exp Brain Res. 2005 Dec;167(3):324-34. doi: 10.1007/s00221-005-0034-x. Epub 2005 Aug 20. PMID 16132974
- [Background] Revel M, Andre-Deshays C, Minguet M. Cervicocephalic kinesthetic sensibility in patients with cervical pain. Arch Phys Med Rehabil. 1991 Apr;72(5):288-91. PMID 2009044
- [Background] Van Den Houte M, Vlemincx E, Franssen M, Van Diest I, Van Oudenhove L, Luminet O. The respiratory occlusion discrimination task: A new paradigm to measure respiratory interoceptive accuracy. Psychophysiology. 2021 Apr;58(4):e13760. doi: 10.1111/psyp.13760. Epub 2021 Jan 12. PMID 33438245
- [Background] Bogaerts K, Walentynowicz M, Van Den Houte M, Constantinou E, Van den Bergh O. The Interoceptive Sensitivity and Attention Questionnaire: Evaluating Aspects of Self-Reported Interoception in Patients With Persistent Somatic Symptoms, Stress-Related Syndromes, and Healthy Controls. Psychosom Med. 2022 Feb-Mar 01;84(2):251-260. doi: 10.1097/PSY.0000000000001038. PMID 34840287
- [Background] Vlemincx E, Walentynowicz M, Zamariola G, Van Oudenhove L, Luminet O. A novel self-report scale of interoception: the three-domain interoceptive sensations questionnaire (THISQ). Psychol Health. 2023 Sep-Oct;38(9):1234-1253. doi: 10.1080/08870446.2021.2009479. Epub 2021 Dec 7. PMID 34875958
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Nijenhuis, E. R. S., van der Hart, O., & Kruger, K. (2002). The psychometric characteristics of the Traumatic Experiernce Checklist (TEC): First findings among psychiatric outpatients. Clinical Psychology & Psychotherapy, 9(3). 200-210. DOI: 10.1002/cpp.332
- [Background] Bagby RM, Parker JD, Taylor GJ. The twenty-item Toronto Alexithymia Scale--I. Item selection and cross-validation of the factor structure. J Psychosom Res. 1994 Jan;38(1):23-32. doi: 10.1016/0022-3999(94)90005-1. PMID 8126686
- [Background] Ramakers I, Fonteyne R, Walentynowicz M, Oudenhove LV, Houte MVD, Bogaerts K. The Need for Controllability and Predictability questionnaire (NCP-q): psychometric properties and preliminary findings in a clinical sample. Health Psychol Rep. 2025 Jan 24;13(2):201-214. doi: 10.5114/hpr/195733. eCollection 2025. PMID 40487476
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Frost, R. O., Marten, P., Lahart, C., & Rosenblate, R. (1990). The dimensions of perfectionism. Cognitive Therapy and Research, 14(5), 449-468. https://doi.org/10.1007/BF01172967
- [Background] Tellegen A, Atkinson G. Openness to absorbing and self-altering experiences ("absorption"), a trait related to hypnotic susceptibility. J Abnorm Psychol. 1974 Jun;83(3):268-77. doi: 10.1037/h0036681. No abstract available. PMID 4844914
- [Background] Overbeek, T., Schrueurs, K., & Griez, E. (1999). MINI-the international neuropsychiatric interview. Dutch version 5.0.0 DSM-IV. Maastricht (Netherlands): University of Maastricht.